CLINICAL TRIAL: NCT02716597
Title: Effect of Albumin Administration on Vasopressor Duration in Resolving Septic Shock
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: difficulty enrolling
Sponsor: Alexander Flannery, 859-323-4011 (Other)
Responsible Party: Sponsor-Investigator, Alexander Flannery, 859-323-4011, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 14-0727-F2L
Record Dates: First submitted 2016-02-19; First posted 2016-03-23 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Shock, Septic
Keywords: albumin, septic shock
MeSH Terms: conditions — Shock, Septic | interventions — Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

ARMS (2):
- 25% Albumin (Experimental): 25% albumin 75 grams IV over 1 hour once.
  Interventions: Drug: 25% Albumin
- Placebo (Placebo Comparator): 0.9% normal saline 200mL IV over 1 hour once.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 25% Albumin
  Arms: 25% Albumin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The role of albumin in sepsis has been controversial for decades. Although hypoalbuminemia has been associated with worse outcomes in sepsis, definitive evidence does not exist that replacing albumin in these patients improves outcomes. However, subgroup analyses from large clinical trials indicate that albumin may reduce mortality in septic shock, and in particular, may reduce the time a patient requires vasopressor support. Given this background, we are conducting this study to evaluate the role of albumin replacement in the patient with resolving septic shock to determine if albumin administration reduces the time a patient requires vasopressor support, reduces the time required for central line, and ultimately whether any potential benefit in terms of reduction of vasopressor support is associated with ICU length of stay and other outcomes. The approach is unique from larger trials of albumin in that it is a septic shock study geared at a particular phenotype of the patient in septic shock and evaluating a specific intervention at a specific time point in the course of septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older who meet the clinical criteria for septic shock

   a. Presence of two or more of the following: i. A core temp ≥38C or ≤36C; ii. A heart rate ≥90 beats/min; iii. A respiratory rate ≥ 20 breaths/min or PaCO2 ≤32mmHg or use of mechanical ventilation for an acute process; iv. A white blood cell count ≥12000/ml or ≤4000/ml or immature neutrophils > 10%.

   b. Presence of defined (or suspected) site of infection as show by at least one of the following criteria: i. An organism grown in blood or sterile site; ii. An abscess or portion of infected tissue; iii. Suspected infection despite culture growth by the attending physician. c. Infusion of vasopressors is required to maintain blood pressure
2. Vasopressor requirements

   a. Patients can be considered for study inclusion when his/her vasopressor requirements are as follows: i. Norepinephrine 0.04-0.25 mcg/kg/min (plus or minus vasopressin) OR phenylephrine 0.2-2 mcg/kg/min (plus or minus vasopressin) AND ii. Last measured lactate value was < 4 mmol/L AND iii. The patient is on stable or decreasing doses of vasopressors for 8 hours or more. This 8 hour measurement will start at the maximum amount of vasopressor support within the range defined in i. above.
3. Serum albumin level <2.5g/dl. The level must be drawn within the last 24 hours of Time=0.

Exclusion Criteria:

1. Patients <18 years old
2. Albumin administration 24 hours prior to the time of enrollment (Time=0)
3. Prisoners
4. Terminal state
5. Known adverse reaction to albumin administration
6. Pregnancy
7. Pathological conditions in which albumin administration is clinically indicated (hepatic cirrhosis with ascites, hepatorenal syndrome, intestinal malabsorption syndrome, nephrotic syndrome, burns)
8. Patients with acute liver failure or cirrhosis
9. Patients on continuous renal replacement therapy
10. Patients who are morbidly obese ≥40kg/m2
11. Religious objection to the administration of human blood products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Time to Cessation of Vasopressor Therapy | Until ICU Discharge (up to 28 days after study drug administration)
  Time from study drug administration to when the patient no longer requires vasopressor support

SECONDARY OUTCOMES:
Time to Central Line Discontinuation | Until ICU Discharge (up to 28 days after study drug administration)
  Time from study drug administration to discontinuation of a patient's central line
Time on Mechanical Ventilation | Until ICU Discharge (up to 28 days after study drug administration)
  Time the patient requires mechanical ventilation during their ICU stay
ICU Mortality | Until ICU Discharge (up to 28 days after study drug administration)
ICU Length of Stay | Until ICU Discharge (up to 28 days after study drug administration)
  How long the patient is in the intensive care unit
Central venous pressure | Measured hourly until 24 hours following study drug administration
  The central venous pressure (in mm Hg) will be measured hourly from a central line until 24 hours following study drug administration.
Heart Rate | Measured hourly until 24 hours following study drug administration
  The heart rate will be measured hourly until 24 hours following study drug administration.
Mean arterial pressure | Measured hourly until 24 hours following study drug administration
  The mean arterial pressure (in mm Hg) will be measured hourly from an arterial line until 24 hours following study drug administration.
Serum creatinine | Measured the day following study drug administration
  Serum creatinine will be measured with AM labs the day following study drug administration and compared with baseline.
Urine output | Measured for 24 hours following study drug administration
  Urine output (in mL) will be measured as part of routine care and totaled for the 24 hour urine output since study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander H. Flannery, Pharm.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky HealthCare Chandler Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No